CLINICAL TRIAL: NCT03284879
Title: OTEZLA® Tablets Drug Use-Results Survey
Brief Title: Post-Marketing Surveillance Study of OTEZLA
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-10004-PSOR-018
Record Dates: First submitted 2017-08-31; First posted 2017-09-15 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis
Keywords: Psoriasis vulgaris; Psoriasis arthropathica; Serious infections; Gastrointestinal Disorders; Serious Hypersensitivity; Weight Decrease; Vasculitis; Malignancies; Depression and Suicidal Ideation
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic; Gastrointestinal Diseases; Weight Loss; Vasculitis; Neoplasms; Depression; Suicidal Ideation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with PsV and PsA treated with OTEZLA Tablets: Patients with psoriasis vulgaris and patients with psoriatic arthritis who are treated with OTEZLA Tablets

SUMMARY:
To evaluate the safety and efficacy of OTEZLA in actual clinical settings of use in patients with Psoriasis vulgaris that is with an inadequate response to topical therapies and Psoriasis arthropathica

1. Planned registration period 2 years
2. Planned surveillance period for 4 years from 6 months after launch

ELIGIBILITY:
Inclusion Criteria:

- Patients who have received a diagnosis of either of the following diseases and have received OTEZLA for the first time will be included in this survey.

* Psoriasis vulgaris that is with an inadequate response to topical therapies
* Psoriasis arthropathica

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have received a diagnosis of either of the following diseases and have received OTEZLA for the first time will be included in this survey.
  * Psoriasis vulgaris that is with an inadequate response to topical therapies
  * Psoriasis arthropathica
Sampling Method: Probability Sample
Enrollment: 1086 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to approximately 12 months
  Number of participants with adverse events
General Improvement Rating | Approximately 1 year from administration
  General Improvement Rating will be assessed by physician's observation
General health assessment on VAS | Approximately 1 year from administration
  Visual Analog Scale (VAS) pain will be used for psoriatic arthritis patients' assessment.
Changes in physician general assessment | Approximately 1 year from administration
  PGA: assessment for psoriatic vulgaris by physician to classify disease activity in a consistent manner
Percentage of patients with Dermatology Life Quality Index (DLQI) | Approximately 1 year from administration
  The Dermatology Life Quality Index or DLQI is a dermatology-specific Quality of Life instrument. It is a simple 10-question validated questionnaire
Change from baseline activity for arthritis | Approximately 1 year from administration
  Activity for arthritis Baseline is calculated by Disease Activity Score-DAS28 method

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Tugi dermatology clinic, Kitakyushu, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Ohtsuki M, Okubo Y, Saeki H, Igarashi A, Imafuku S, Abe M, Chaudhari S, Yaguchi M, Emoto A, Morita A. Safety and effectiveness of apremilast in Japanese patients with psoriatic disease: Results of a post-marketing surveillance study. J Dermatol. 2024 Jul;51(7):950-963. doi: 10.1111/1346-8138.17270. Epub 2024 May 22. PMID 38775204
- [Background] Ohtsuki M, Okubo Y, Saeki H, Igarashi A, Imafuku S, Abe M, Saito K, Ogawa R, Morita A. Clinical Characteristics and Safety Profiles of Japanese Psoriasis Patients Who Continued Apremilast Treatment for 6 and 12 Months: A Post Hoc Analysis of an Apremilast Postmarketing Surveillance Study. J Dermatol. 2025 Jun;52(6):1059-1065. doi: 10.1111/1346-8138.17764. Epub 2025 May 10. PMID 40346955
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Expanded Access for CC-10004 — https://clinicaltrials.gov/ct2/show/NCT03284879?term=CC-10004-PSOR-018&rank=1